CLINICAL TRIAL: NCT04862819
Title: Clinical, Biochemical and Microbiological Evaluation of a New Local Drug Delivery in the Nonsurgical Treatment of Periodontitis
Brief Title: Evaluation of a New Local Drug Delivery in the Nonsurgical Treatment of Periodontitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: KB776-2019
Record Dates: First submitted 2021-03-02; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-01

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- scaling root planning (Active Comparator): patients in this group will have a scaling root planing procedure only
  Interventions: Procedure: scaling root planing
- scaling root planning with new local drug delivery (Experimental): patients in this group will have a scaling root planing procedure and a drug administered
  Interventions: Drug: new local drug delivery; Procedure: scaling root planing

INTERVENTIONS:
Drug: new local drug delivery — In the first group, on one side of the dental arch, the drug under evaluation will be used, and on the other side srp
  Other Names: New LDD
  Arms: scaling root planning with new local drug delivery
Procedure: scaling root planing — In the second group, on one side of the dental arch srp will be performed
  Other Names: Scaling root planing (gold standard treatment)

SUMMARY:
The aim of the planned randomized clinical trial will be the clinical and microbiological evaluation of the new intracellular drug developed in cooperation with the Chair and Department of Drug Form Technology of the Medical University and the Department and Department of Pharmaceutical Microbiology and Parasitology of the Medical University in Wrocław.

DETAILED DESCRIPTION:
Clinical trials will be conducted on 60 patients of the Department of Periodontology of the Medical University of Wrocław with 3rd or 4th degree generalized periodontitis, who will consent to participate in the research by signing the documentation approved by the Bioethics Committee of our University. The exclusion criteria will be: the presence of general diseases affecting the clinical condition of the periodontium, hypersensitivity to the drug used in the carrier system, lack of proper oral hygiene, active nicotinism and age over 65 years. The research will be carried out according to the scheme of parallel randomization and double-blinded trial in two groups of 30 people. All qualified patients will undergo an initial period of periodontal treatment and scaling / root planning.

In the first group, on one side of the dental arch, the drug under evaluation will be used, and on the other side, placebo with a change of side in every second patient. In the other group, the drug under evaluation or placebo will be used on one side, and the SRP treatment with alternation of sides on the other side for every second patient.

ELIGIBILITY:
Inclusion Criteria:

* stage- 3rd degree generalized periodontitis
* stage 4th degree generalized periodontitis

Exclusion Criteria:

* presence of general diseases affecting the clinical condition of the periodontium,
* hypersensitivity to the drug used in the carrier system,
* lack of proper oral hygiene
* active nicotinism
* age over 65 years

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-02 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
changes in PD (pocket depth in millimetres ) | 3 month
  Change in depth of periodontal pockets measured from the bottom of the pocket to the edge of the gum in millimetres using periodontal probe
changes in CAL (clinical attachment level in millimetres ) | 3 month
  Change in clinical attachment level of periodontal pockets measured from the Cement-enamel junction to the bottom of the pocket in millimetres using periodontal probe
changes in microbiome (rt PCR test) | 3 month
  change in microbiological and biochemical parameters of pocket microbiome using PCR real time test 3 months after Local dryg delivery (LDD) application( taken from the gingival pocket with gingival fluid with a paper filter. There will be six bacterial strains and the bacterial total load assessed)

CONTACTS AND LOCATIONS:
Overall Officials: Małgorzata Szulc, phd, Study Director — wroclaw medical univeristy; Tomasz Konopka, prof, Principal Investigator — wroclaw medical univeristy
Locations (2):
- Poland (2):
  - Jacek Zborowski, Wroclaw, Lower Silesian Voivodeship
  - Wroclaw Medical University, Wroclaw

IPD SHARING:
Plan to Share IPD: No